CLINICAL TRIAL: NCT04138914
Title: Phase II Trial of Focal Cryotherapy for Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2482
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Focal Cryotherapy (Experimental): Focal Cryotherapy using 2 freeze-thaw cycles
  Interventions: Device: Focal Cryotherapy

INTERVENTIONS:
Device: Focal Cryotherapy — Ablation of the cancer focus within the prostate using cryotherapy
  Other Names: Focal Therapy; Focal Cryoablation

SUMMARY:
The current standard of care treatment for prostate cancer confined to the prostate is surgical removal or irradiation of the entire prostate gland. This is effective at curing cancer but result in damage to critical adjacent structures such as the urinary sphincter muscle and erectile nerves resulting in impaired urinary continence and erectile dysfunction. The concept of focal therapy is to treat just the dangerous focus of cancer in the prostate while monitoring the rest of the gland, thus avoiding impairment of urinary continence and erectile function. We aim to evaluate the degree of preservation of continence and erectile function and early oncological outcomes in patients undergoing focal therapy of the prostate using cold energy or cryo- ablation. In this study, we seek to evaluate patient reported outcomes in urinary, sexual, bowel and general health areas at fixed time points after focal cryo-ablation in selected patients with low-volume, localized cancer. The primary goal of this study is to demonstrate whether there is a deterioration of scores in these health areas over 1 year of follow-up. The secondary goal is to measure cancer control at 1 year re-biopsy. Further goals include longer follow-up to monitor cancer progression rates and impact on patient survival.

ELIGIBILITY:
Inclusion criteria:

* PSA (prostate specific antigen) ≤ 20
* Biopsy Gleason score ≤ 4+4
* mpMRI shows no gross extracapsular extension
* mpMRI shows index lesion volume < 3 ml
* ≤ 2 biopsy confirmed lesions on mpMRI

Exclusion criteria:

* American Society of Anesthesiologist score >3
* Very high grade cancer (Gleason score > 4+4)
* >2 index lesions
* Multifocal cancer (any other Gleason >3+3 present and/or Gleason 3+3 at > 3 biopsy cores at another site) - Not eligible for mpMRI
* Not fit for robotic transperineal saturation biopsy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2041-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in EPIC (Expanded Prostate Composite Index) subdomain score at 1, 3, 6, 12 months compared to baseline | 1,3,6 and 12 months
Number of Participants with Treatment-Related Adverse Events assessed by the Clavien-Dindo Scale | at 3 months

SECONDARY OUTCOMES:
Infield (focally treated area) and Outfield (untreated area) positive biopsy rate at 12 months | at 12 months

OTHER OUTCOMES:
Local Progression Rate as measured by follow-up mpMRI (multi parametric magnetic resonance imaging) | up to 10 years
Metastatic Rate as measured by Bone Scan, CT or mpMRI | up to 10 years
Death Rate | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kae Jack Tay, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tay KJ, Scheltema MJ, Ahmed HU, Barret E, Coleman JA, Dominguez-Escrig J, Ghai S, Huang J, Jones JS, Klotz LH, Robertson CN, Sanchez-Salas R, Scionti S, Sivaraman A, de la Rosette J, Polascik TJ. Patient selection for prostate focal therapy in the era of active surveillance: an International Delphi Consensus Project. Prostate Cancer Prostatic Dis. 2017 Sep;20(3):294-299. doi: 10.1038/pcan.2017.8. Epub 2017 Mar 28. PMID 28349978
- [Background] Tay KJ, Polascik TJ, Elshafei A, Tsivian E, Jones JS. Propensity Score-Matched Comparison of Partial to Whole-Gland Cryotherapy for Intermediate-Risk Prostate Cancer: An Analysis of the Cryo On-Line Data Registry Data. J Endourol. 2017 Jun;31(6):564-571. doi: 10.1089/end.2016.0830. PMID 28385075
- [Background] Tay KJ, Cheng CWS, Lau WKO, Khoo J, Thng CH, Kwek JW. Focal Therapy for Prostate Cancer with In-Bore MR-guided Focused Ultrasound: Two-Year Follow-up of a Phase I Trial-Complications and Functional Outcomes. Radiology. 2017 Nov;285(2):620-628. doi: 10.1148/radiol.2017161650. Epub 2017 Jun 26. PMID 28654336
- [Background] Tay KJ, Amin MB, Ghai S, Jimenez RE, Kench JG, Klotz L, Montironi R, Muto S, Rastinehad AR, Turkbey B, Villers A, Polascik TJ. Surveillance after prostate focal therapy. World J Urol. 2019 Mar;37(3):397-407. doi: 10.1007/s00345-018-2363-y. Epub 2018 Jun 9. PMID 29948045
- [Background] Bahn D, de Castro Abreu AL, Gill IS, Hung AJ, Silverman P, Gross ME, Lieskovsky G, Ukimura O. Focal cryotherapy for clinically unilateral, low-intermediate risk prostate cancer in 73 men with a median follow-up of 3.7 years. Eur Urol. 2012 Jul;62(1):55-63. doi: 10.1016/j.eururo.2012.03.006. Epub 2012 Mar 21. PMID 22445223
- [Derived] Tan YG, Law YM, Ngo NT, Khor LY, Tan PH, Ong EHW, Yuen JSP, Ho HSS, Tuan JKL, Kanesvaran R, Gupta RT, Rozen S, Chua MLK, Polascik TJ, Tay KJ. Patient-reported functional outcomes and oncological control after primary focal cryotherapy for clinically significant prostate cancer: A Phase II mandatory biopsy-monitored study. Prostate. 2023 Jun;83(8):781-791. doi: 10.1002/pros.24517. Epub 2023 Mar 9. PMID 36895163